CLINICAL TRIAL: NCT03175263
Title: OnabotulinumtoxinA Injections in Chronic Migraine, Targeted to Sites of Pericranial Myofascial Pain : an Observational, Open Label, Real-life Cohort Study.
Brief Title: OnabotulinumtoxinA Injections in Chronic Migraine, Targeted to Sites of Pericranial Myofascial Pain
Status: Completed | Type: Observational
Sponsor: University Hospital, Limoges (Other)
Responsible Party: Sponsor
Other Study IDs: I17022
Record Dates: First submitted 2017-06-01; First posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Chronic Migraine
Keywords: onabotulinumtoxinA, chronic migraine, myofascial pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with chronic migraine: Patients with chronic migraine refractory to conventional treatments

SUMMARY:
This study was an observational, open-label, cohort-study conducted in accordance with the principles of the Helsinki Declaration. We prospectively and systematically recorded data from the patients and analyzed them retrospectively. During a first phase, called adaptation period, the injector (DR) used a follow-the-pain approach in order to determine the optimal injection scheme for each individual. The possible injection sites were the corrugator, temporalis, and trapezius muscles. Patients were systematically asked about the usual topography and time course of migraine attacks, and the existence of pain or stiffness of the cervical muscles. If the pain was predominantly located in the frontotemporal area, the corrugator and temporalis muscles were injected bilaterally. When the patients had predominant pain in the back of the head, or when their headache pain frequently started and/or ended in the trapezius muscles, both trapezius muscles were injected. These muscle groups were injected together if pain was both frontotemporal and cervico-occipital. When this first set of injections was efficacious, patients were re-injected in the same manner at the time when the frequency of headache days definitely increased. In the absence of efficacy, the paradigm was modified using the same follow-the-pain approach. Once the best procedure was determined for each patient, it was reproduced at each subsequent injection session. This adaptation phase could necessitate up to three sessions. The observation period started 8 weeks before the first efficacious injection and ended 2 months after the second consecutive efficacious injection, or in case of inefficacy. Throughout the adaptation and the observation phases, patients kept a headache diary where they were asked to note the days with headache and the use of rescue medication.

ELIGIBILITY:
Inclusion Criteria:

* Patients refractory to conventional treatments

Exclusion Criteria:

* Contra-indication to botulinum toxin treatment Inability to sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic migraine
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2008-09-01 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
frequency of headache days | Week 8
  change from baseline in frequency of headache days (as recorded in the patient diary) for the 2 months-period ending with week 8

SECONDARY OUTCOMES:
the proportion of patients with a ≥ 70% decrease in headache day frequency | Week 8
  the proportion of patients with a ≥ 70% decrease in headache day frequency
the decrease in triptan consumption | Week 8
  the decrease in triptan consumption
the assessment of patient satisfaction | Week 8
  the assessment of patient satisfaction on a 0 to10 numerical scale (0=no improvement, and 10=maximum possible improvement).

CONTACTS AND LOCATIONS:
Overall Officials: Daniele RANOUX, PH, Principal Investigator — University Hospital, Limoges

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ranoux D, Martine G, Espagne-Dubreuilh G, Amilhaud-Bordier M, Caire F, Magy L. OnabotulinumtoxinA injections in chronic migraine, targeted to sites of pericranial myofascial pain: an observational, open label, real-life cohort study. J Headache Pain. 2017 Dec;18(1):75. doi: 10.1186/s10194-017-0781-7. Epub 2017 Jul 21. PMID 28733943